CLINICAL TRIAL: NCT04170920
Title: Pilot Study of a Mobile Health Strategy to Improve Medication Adherence in Breast Cancer Survivors Receiving Aromatase Inhibitors
Brief Title: Pilot Study of a an App to Improve Medication Adherence in Breast Cancer Survivors Receiving AIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tarah J Ballinger, MD, Assistant Professor of Clinical Medicine, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CTO-IUSCC-0715
Record Dates: First submitted 2019-11-13; First posted 2019-11-20 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer; DCIS
Keywords: breast cancer; DCIS; aromatase inhibitor
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mobile Health Application Intervention (Experimental): LifeExtend-AI (LX-AI) will be piloted by adding Aromatase Inhibitor (AI)- specific features to LifeExtend, an already existing healthy lifestyle behavior application produced by LifeOmic. This application includes features for tracking activity, diet, sleep, and body weight, as well as creating "to-do" lists and participating in closed social networking for support and encouragement. LifeExtend-AI will add features to track AI adherence and patient-reported joint pain, with alerts sent to both the participant and the healthcare team in response to these parameters. In addition, the app contains educational videos and articles, to which articles addressing management of AI- related toxicities (including exercise) will be added.
  Interventions: Device: LifeExtend-AI

INTERVENTIONS:
Device: LifeExtend-AI — LifeExtend-AI (LX-AI) will be piloted by adding AI- specific features to LifeExtend, an already existing healthy lifestyle behavior application produced by LifeOmic. This application includes features for tracking activity, diet, sleep, and body weight, as well as creating "to-do" lists and participating in closed social networking for support and encouragement. LifeExtend-AI will add features to track AI adherence and patient-reported joint pain, with alerts sent to both the participant and the healthcare team in response to these parameters. In addition, the app contains educational videos and articles, to which articles addressing management of AI- related toxicities (including exercise) will be added.

SUMMARY:
The purpose of this study is to evaluate the feasibility of an mobile-health strategy to improve patient-reported symptoms, promote life-saving medication adherence, and encourage healthy lifestyle behaviors in early stage breast cancer survivors receiving adjuvant Aromatase inhibitors, while beginning to predict psycho-social and demographic characteristics of those who benefit most from this approach. This will provide preliminary experience and evidence for larger, randomized clinical trials evaluating this methodology, which will have immediate and scalable influence on cancer survivor ship.

DETAILED DESCRIPTION:
This is a single arm, prospective, observational study enrolling up to 50 patients to the intervention in groups of 10 within Indiana University Simon Cancer Center. Subjects must meet eligibility at the time of informed consent. Once 10 eligible subjects are identified and have signed informed consent, each subject will return for their baseline visit and begin the app intervention with their group of 10.

Primary Objective Evaluate the feasibility of a smartphone application, LifeExtend-AI, in patients with early stage breast cancer currently prescribed aromatase inhibitor therapy, determined by patient usage of the application.

Secondary Objectives

1. Determine a preliminary estimate of effect size of the app intervention on medication adherence, by self- report using the Brief Medication Questionnaire
2. Determine a preliminary estimate of effect size of the app intervention on patient -reported AI arthralgia, as measured by the Basic Pain Inventory (BPI).
3. Determine a preliminary estimate of effect size of the app intervention on patient reported health associated quality of life, measured by the Functional Assessment of Cancer Therapy- Endocrine symptoms (FACT-ES) questionnaire.
4. Determine a preliminary estimate of the effect size of the app intervention on patient satisfaction with healthcare team communication, measured by the FACIT- Treatment Satisfaction-Patient Satisfaction questionnaire (FACIT-TS-PS).
5. Determine a preliminary estimate of effect size of the app intervention on patient reported health depression and anxiety, as measured by the Hospital Anxiety and Depression Scale (HADS).
6. Determine a preliminary estimate of effect size of the app intervention on patient reported physical activity level, as measured by the International Physical Activity Questionnaire (IPAQ).
7. Investigate psychosocial and behavioral determinants of application usage and subsequent medication adherence, including perceived AI necessity, fear of cancer recurrence, health self-efficacy, and e-health literacy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old at the time of informed consent
2. Regular access to a smartphone capable of downloading the application

   1. iOS 11 or later (iPhone5, iPhone SE or newer)
   2. Android 6 or later (Android 9 is current version)
3. History of DCIS, stage I, II, or III invasive breast cancer
4. Currently prescribed an aromatase inhibitor (letrozole, anastrozole, exemestane) or planned to be initiated on one by the time of signing informed consent. Patient already on an AI must have been prescribed this medication for a total of 36 months or less.

   1. Ovarian suppression with AI is allowed in premenopausal patients.
   2. Prior SERM and now switching to an AI for the first time is allowed.
   3. Concurrent trastuzumab, pertuzumab, or TDM1 is allowed.
   4. Concurrent neratinib or other oral cancer directed medication is not allowed.
5. ECOG performance status of 0-2

Exclusion Criteria:

1. Metastatic breast cancer or other active malignancy

   1. Locally recurrent breast cancer is allowed if treated with surgical excision and AI is prescribed with curative intent.
   2. History of prior treated malignancies, other than breast cancer, that are now stable, are in remission, and do not require active therapy, are acceptable
2. Unable to read the English language or otherwise participate in the study procedures in the opinion of the treating investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Participants who use the LifeExtend-AI application 5 or more days per week | 12 weeks
  Feasibility will be measured by participants who use the application 5 or more days per week

SECONDARY OUTCOMES:
Mean medication adherence using the Brief Medication Questionnaire (BMQ) | Baseline and post intervention (an average of 12 weeks)
  Self report tool for monitoring medication adherence, measuring medication knowledge, beliefs, and recall. A score of 1 or more in each section is a positive screen for non-adherence ,belief barriers, or recall barriers.
Mean pain score of self -reported aromatase inhibitor arthralgia using the Basic Pain Inventory (BPI) | Baseline and post intervention (an average of 12 weeks)
  Mean score of the 9 item scale.
Mean quality of life score, measured by the Functional Assessment of Cancer Therapy- Endocrine symptoms (FACT-ES) | Baseline and post intervention (an average of 12 weeks)
  Likert-scaled questionnaire, with response scores ranging from 0 to 4.
Mean satisfaction with healthcare team communication, measured by the FACIT- Treatment Satisfaction-Patient Satisfaction questionnaire (FACIT-TS-PS) | Baseline and post intervention (an average of 12 weeks)
  Likert-scaled questionnaire, with response scores ranging from 0 to 3.
Mean quality of life, as measured by the Hospital Anxiety and Depression Scale (HADS) | Baseline and post intervention (an average of 12 weeks)
  Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. The HADS uses a scale and therefore the data returned from the HADS is ordinal.
Mean quality of life, as measured by the International Physical Activity Questionnaire (IPAQ) | Baseline and post intervention (an average of 12 weeks)
  MET-min per week: MET level x minutes of activity x events per week. To calculate MET minutes a week multiply the MET value given by the minutes the activity was carried out and again by the number of days that that activity was undertaken.
Mean quality of life, as measured by the eHEALTH literacy scale (ehEALS) | Baseline and post intervention (an average of 12 weeks)
  he eHEALS contains 8 items, measured with a 5-point Likert scale with response options ranging from "strongly disagree" to "strongly agree." Total scores of the eHEALS are summed to range from 8 to 40, with higher scores representing higher self-perceived eHealth literacy.
Mean quality of life, as measured by the Patient Activation Measure (PAM) | Baseline and post intervention (an average of 12 weeks)
  A 13-item survey that assesses a person's underlying knowledge, skills and confidence integral to managing his or herown health and healthcare on a 100 point scale.
Mean quality of life, as measured by the assessment of cancer worry in aromatase inhibitor users | Baseline and post intervention (an average of 12 weeks)
  Mean score of 3 item scale with responses on a 1-10 scale where 0 indicates "not at all" and 10 indicates "a great deal"

CONTACTS AND LOCATIONS:
Overall Officials: Tarah Ballinger, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Melvin & Bren Simon Cancer Center, Indianapolis, Indiana, United States